CLINICAL TRIAL: NCT07380204
Title: In Vivo Quantification of Hsp90 in the Human Brain in Healthy Aging and Neurodegeneration Using the Novel PET Radioligand [11C]HSP990
Brief Title: Quantification of Hsp90 in the Human Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: S68531; 2023-510532-36-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-05; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD); Alzheimer's Disease (AD); Amyotrophic Lateral Sclerosis (ALS)
Keywords: HSP90; PET; test-retest; dosimetry; Parkinson; Alzheimer; ALS
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1: Biodistribution and dosimetry (Experimental): In this part of the study, three healthy volunteers (2 male / 1 female, aged 18-55 years) will undergo consecutive whole-body PET/CT scans over a period of 120 minutes to measure the biodistribution in the body and the radiation exposure of [¹¹C]HSP990 in humans.
  Interventions: Other: [11C]HSP990 PET dosimetry
- 2: Kinetics and variability in the brain (Experimental): In this part of the study, five young healthy volunteers (male/female, aged 18-40 years) will undergo a PET/CT brain scan with a total duration of 120 minutes (70 minutes of scanning - 20 minutes break - 30 minutes scanning). During the scan, the amount of tracer reaching the brain via the bloodstream will be determined using blood samples taken from an artery. In addition, the breakdown of the tracer by the liver and the formation of by-products ("metabolite" analysis) will be measured in order to determine how much intact tracer reaches the brain. This is necessary to quantify the amount of Hsp90 protein in the brain based on the tracer concentration.
  If possible, a simplified approach will be developed to minimize the physical burden of the study for participants in Part 3 of the study.
  All five volunteers will also undergo a retest scan within an interval of one week in order to determine the precision (test-retest reliability).
  Interventions: Other: [11C]HSP990 PET test-retest
- 3: Comparison with patient group (Experimental): In this part of the study, 30 patients (10 with Parkinson's disease [PD], 10 with Alzheimer's disease [AD], and 10 with amyotrophic lateral sclerosis [ALS]) and 10 healthy controls will undergo a dynamic simultaneous PET/CT brain scan, using the least invasive protocol as established in Part 2, to investigate whether the (regional) brain uptake of the tracer [¹¹C]HSP990 differs between healthy aging and patients with neurodegenerative disease.
  Interventions: Other: [11C]HSP990 simplified scan protocol

INTERVENTIONS:
Other: [11C]HSP990 PET dosimetry — 120 minute whole body PET/CT scan with [11C]HSP990 radiotracer
  Arms: 1: Biodistribution and dosimetry
Other: [11C]HSP990 PET test-retest — 2 120-minute brain PET scan with [11C]HSP990 radiotracer
  Arms: 2: Kinetics and variability in the brain
Other: [11C]HSP990 simplified scan protocol — Simplified quantitative [11C]HSP990 PET scan as will be determined in part 2.
  Arms: 3: Comparison with patient group

SUMMARY:
This study tests the radiolabeled molecule ("tracer"), [¹¹C]HSP990, using positron emission tomography (PET) imaging to assess whether it can be used to measure levels of Heat Shock Protein 90 (Hsp90). The protein Hsp90 plays an important role in how proteins in the brain fold into their three-dimensional structure and how this protein helps maintain cellular homeostasis. Since neurodegenerative diseases such as Alzheimer's disease (AD), Parkinson's disease (PD), and amyotrophic lateral sclerosis (ALS) are characterized by disrupted three-dimensional protein folding resulting in protein aggregation, we also aim to measure Hsp90 levels in patients with these conditions.

[¹¹C]HSP990 is a promising tracer for this purpose and has already been extensively tested in animal models with safe and favorable results. The investigator now aims to evaluate this tracer in the human brain in healthy volunteers as well as in patients with Parkinson's disease, Alzheimer's disease and amyotrophic lateral sclerosis. The investigator expects that Hsp90 protein levels will be present at reduced concentrations in patients, possibly in different brain regions depending on the distribution of the disease-causing proteins associated with these disorders.

Since the discovery of the important role of Hsp90 in neurodegenerative diseases, several candidate drugs targeting Hsp90 have been developed in recent years. The imaging method used in this study may support the development of Hsp90-targeting medications by enabling measurement of Hsp90 levels in the brain and assessment of the effects of these drugs.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
* Male or female subjects, age between 18-55 (Part 1, n = 3), 18-40 (Part II, n = 5) or 40-70 (Part III, 40-55 n = 5, 55-70 n = 5) years old.
* Subject is judged to be in good health by the investigator on the basis of medical history, physical examination including vital signs, clinical laboratory test and urinalysis.
* No history or evidence of current major neurological, internal or psychiatric disorder, based on the medical assessment as described hereabove and neuropsychological assessment (SCL-90).
* (Part II and III only: ) In subjects < 60 years of age, a normal structural MRI scan as assessed by expert radiologist. In subjects >= 60 years of age white matter hyperintensities corresponding to a white matter lesion (WML) Fazekas score < 2 on the Age-Related White Matter changes scale are acceptable

Parkinson's disease

* Age 45-85 years.
* Patient has clinically established PD based on the Movement Disorder Society (MDS) diagnostic criteria and is in Hoehn-Yahr stage I-III in the "on" medication state
* Patient has had a previous abnormal DaT-scan confirming the clinical diagnosis.
* Patient is able to understand the patient information brochure and give written informed consent

Alzheimer's disease

* Age 45-85 years.
* MoCA score < 26
* Patient has a diagnosis of probable AD with evidence of the AD pathophysiological process (amyloid PET scan or CSF determination) according to the consensus criteria [McKahn et al 2011, Alzh Dement].
* Patient is able to understand the patient information brochure and give written informed consent.

Amyotrophic lateral sclerosis

* Age 20-85 years.
* Subjects will be recruited at the Neurology department of University Hospitals Leuven and must meet revised El Escorial Criteria and Awaji-Shima criteria for at least possible ALS.
* Patient is able to understand the patient information brochure and give written informed consent.

Exclusion Criteria:

Healthy controls

* Participant has a history of any major disease that may interfere with the investigations or make the subject unfit for participation according to the interpretation by the investigator (especially diabetes mellitus, heart disease, liver and kidney disease, or most forms of cancer).
* Any prior or concomitant treatment(s) that might jeopardise the participant's safety or that would compromise the integrity of the Trial .
* Participation in an interventional Trial with an investigational medicinal product (IMP) or device.
* Evidence of cognitive impairment.
* Subject has a history or evidence of psychiatric disease.
* Subject has renal impairment with eGFR < 60 ml/min.
* Subject is currently a user (including ''recreational use'') of any illicit drugs, including cannabis, or has a history of drug or alcohol abuse.
* (Part II and III only: ) Subject has a contra-indication for MRI scanning.
* Subject has a known hypersensitivity to any of the excipients that are present in the radiopharmaceutical preparations or to any of the excipients listed in the IMPD for [11C]HSP990.
* Subject suffers from claustrophobia or cannot tolerate confinement during PET-MRI scanning procedures. Subject cannot lie still for at least 70 minutes inside a scanner.
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e., weightlifting, running, bicycling) from the time of the pre-study visit until the end of scanning;
* Subject does not understand the study procedures.
* Subject is unwilling or unable to perform all of the study procedures or is considered unsuitable in any way by the principal investigator.
* Subject is pregnant (according to Ulti Med hCG urine test) or is breastfeeding.
* Subject is a woman of childbearing potential who does not agree to apply appropriate contraception methods during study participation and continues to do so for at least 6 months after study completion. For WOCBP: contraception methods with a relatively high Pearl index (natural methods, minipill outside postpartum period, spermicides or condoms in monocontraception or no usage of contraception when sexually active) are not accepted.
* Subject is a man with a pregnant or non-pregnant WOCBP partner, who does not agree to use a condom and continue to do so until 90 days after study completion. In addition, the non-pregnant WOCBP partner should use a highly effective method of contraception.
* Subject does not agree that incidental findings are communicated to the general practitioner and to the participant him/herself.
* (Part II and III only: ) An abnormal Allen test or hypersensitivity/allergy to lidocaine.
* (Part II and III only: ) Anticoagulant therapy is an exclusion criterium for undergoing arterial sampling as part of the study. Subjects that have anticoagulant therapy can participate in the study parts without arterial sampling.

Parkinson's disease:

* Neuropsychiatric diseases other than the cohort inclusion condition
* Major internal medical comorbidity, in particular diabetes or heart disease
* Subject has renal impairment with eGFR < 60 ml/min.
* White matter lesion load on FLAIR Fazekas score 2 or higher or other relevant MRI abnormalities
* History of alcohol abuse or current alcohol abuse (chronic use of more than 15 units per week) or drug use
* Contraindications for MR
* Subject has a known hypersensitivity to any of the excipients that are present in the radiopharmaceutical preparations or to any of the excipients listed in the IMPD for [11C]HSP990.
* Subject suffers from claustrophobia or cannot tolerate confinement during PET scanning procedures; subject cannot lie still for 70 minutes inside the scanner.
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e., weightlifting, running, bicycling) from the time of the pre-study visit until the end of scanning.
* Subject does not understand the study procedures or does not have a guardian who understands the study procedures.
* Subject (or guardian) is unwilling or unable to perform all of the study procedures or is considered unsuitable in any way by the principal investigator.
* Subject does not agree that incidental findings are communicated to the general practitioner and to the participant him/herself.
* Subject is pregnant (according to Ulti Med hCG urine test) or breastfeeding.
* Subject is a woman of childbearing potential who does not agree to apply appropriate contraception methods during study participation and continues to do so for at least 6 months after study completion. For WOCBP* : contraception methods with a relatively high Pearl index (natural methods, minipill outside postpartum period, spermicides or condoms in monotherapy or no usage of contraception when sexually active) are not accepted.
* Subject is a man with a pregnant or non-pregnant WOCBP partner, who does not agree to use a condom and continue to do so until 90 days after study completion. In addition, the non-pregnant WOCBP partner should use a highly effective method of contraception.
* Anticoagulant therapy is an exclusion criterium for undergoing arterial sampling as part of the study. Subjects that have anticoagulant therapy can participate in the study parts without arterial sampling.

Alzheimer's disease:

- cf. Parkinson's Disease exclusion criteria

Amytorphic lateral sclerosis:

* cf. Parkinson's Disease exclusion criteria
* Subject has confined upper motor neuron involvement (i.e. primary lateral sclerosis) or confined lower motor neuron involvement (i.e. progressive muscular atrophy).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Quantification of HSP90 in the human brain | This will be assessed right after each scan in cohort 2 and 3. (Estimated visit lenght in cohort 2 will be 4 hours for each scanning procedure. In cohort 3 this will be optimized based on the results of cohort 2.)
  To quantify and compare Hsp90 levels in vivo in the human brain of healthy volunteers and patients with neurodegenerative disorders using the novel PET radioligand [11C]HSP990.

SECONDARY OUTCOMES:
To assess the safety and clinical tolerance of [11C]HSP990 administration. | From enrollment until 1 week after completion of scan.
  The impact of [11C]HSP990 administration on clinical symptoms and signs and biochemistry values will be evaluated. Baseline values will be recorded and subjects will be assessed clinically and with dual biochemical analysis (before PET and after PET). Adverse events will be scored as mild, moderate or severe.
  We hypothise that administration of [11C]HSP990 is safe and in view of the low mass dose (< 10 µg) does not result in significant changes in vitals, clinical assessment or biochemistry, or subjective complaints other than those that may be related to the procedure (e.g., catheter placement).
To determine the radiation dosimetry of [11C]HSP990 in humans. | This will be assessed right after each scan in cohort 1. (Estimated lenght of the scanning visit is 4 hours.)
  Effective doses will be determined. The hypothesis is that in young healthy volunteers administration of [11C]HSP990 results in significant brain uptake and is partially hepatobiliary and renally cleared, and results in an effective dose between 3 to 8 microSv/MBq.
To determine the optimal brain tracer kinetic modelling approach and test-retest variation (TRV) for [11C]HSP990 brain PET in humans. | This will be assessed right after each scan in cohort 2. (Estimated lenght of each scanning visit is 4 hours.)
  Total distribution volume (VT) for [11C]HSP990 will be determined using the arterial brain input and response function. The hypothesis is that [11C]HSP990 PET allows for quantifying total Hsp90 distribution volume in the human brain with a 2TCM as the preferred quantitative approach. VT for [11C]HSP990 re-test scans will be determined and TRV will be calculated. The hypothesis is that the absolute short term test-retest will be acceptable (below 10 %).
To determine the optimal imaging protocol for quantifying Hsp90 levels in human brain using [11C]HSP990 and develop if possible, a simplified imaging protocol or patient comfort. | This will be assessed right after each scan in cohort 2. (Estimated lenght of the scanning visit is 4 hours.)
  It will be assessed if less invasive shorter imaging protocols can lead to equivalent outcome parameters in terms of VT. The hypothesis is that dynamic [11C]HSP990 PET combined with an image-derived input function and venous blood sampling based radiometabolite quantification can be used as a less invasive imaging protocol to quantify Hsp90 levels in human brain. Moreover, a shorter simplified coffeebreak protocol (e.g. 0-50 min p.i. dynamic imaging followed by 20 min break and 20 min dynamic imaging) can be used as a more patient friendly and shorter imaging protocol.
To assess age-dependency of Hsp90 levels in healthy human brain using [11C]HSP990 | This will be assessed right after each scan in cohort 2 and 3. (Estimated visit lenght in cohort 2 will be 4 hours for each scanning procedure. In cohort 3 this will be optimized based on the results of cohort 2.)
  The hypothesis is that compared to young healthy volunteers, [11C]HSP990 availability measured by VT is reduced upon healthy ageing and inversely related to age.
To compare Hsp90 levels in healthy human brain versus patients with neurodegeneration using [11C]HSP990 | This will be assessed right after each scan in cohort 2 and 3. (Estimated visit lenght in cohort 2 will be 4 hours for each scanning procedure. In cohort 3 this will be optimized based on the results of cohort 2.)
  Based on preclinical findings, the hypothesis is that [11C]HSP990 VT in all forms of investigated neurodegeneration is globally lower than age-matched healthy volunteers and disease severity/duration is negatively correlated to the reduction of [11C]HSP990 VT.
To assess the regional brain pattern of [11C]HSP990 PET in neurodegeneration | This will be assessed right after each scan in cohort 3. (Estimated scanning visit lenght in will be 3 hours.)
  The regional pattern of reduced [11C]HSP990 uptake (VT) will be assessed and correlated to DaT-scan in PD and amyloid PET in AD. The hypothesis is that in patients with neurodegeneration [11C]HSP990 VT is predominantly reduced in more affected brain regions.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Laere, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaam-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
To be determined.